CLINICAL TRIAL: NCT06278610
Title: Accuracy of Ultrasound Scan in Patients Undergoing Pelvic Exenteration and Laterally Extended Pelvic Resection
Brief Title: Pelvic Exenteration and Laterally Extended Pelvic Resection
Acronym: Pre-PEX
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3612
Record Dates: First submitted 2023-02-27; First posted 2024-02-26 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Gynecologic Cancer; Surgical Procedure, Unspecified
Keywords: pelvic; resection; exenteration
MeSH Terms: interventions — Diagnostic Tests, Routine; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PELVIC EXENTERATION — PELVIC EXENTERATION
  Other Names: Diagnostic Test: For example, imaging,; Procedure/Surgery

SUMMARY:
Growing evidence in literature is supporting the role of ultrasound scan (US) as accurate tool in diagnosis and staging of gynecologic cancers. In particular, different studies demonstrated the accuracy of US in assessing endometrial, cervical, and ovarian cancer in the primary setting. However, the number of studies investigating the role of US in the recurrent setting is limited. Moreover, there is no evidence in literature exploring the role of US in laterally-extended pelvic recurrences from gynecologic cancer, where the Magnetic Resonance Imaging (MRI) scan is still considered the most accurate tool.

DETAILED DESCRIPTION:
All consecutive patients who are planned to undergo pelvic exenteration or laterally extended pelvic resection at Policlinico Agostino Gemelli IRCCS, will undergo ultrasound scan at the time of the pre-operative anesthetic assessment or the day before the planned surgery. A pre-defined case report form (CRF) will be filled by the ultrasound examiner. The ultrasound characteristics will be compared with the final histology (considered the referral standard).

The ultrasound examinations will be carried out using high-end ultrasound equipment. The frequency of the vaginal probes varied between 5.0 and 9.0 MHz. All examinations will be performed by a specialist obstetrics and gynecology with expertise in gynecologic oncology ultrasound scan. A subjective semi-quantitative assessment of the amount of blood flow within the examined lesion will be made (color score): a score of 1 was recorded when no blood flow could be found; 2 when only minimal/moderate flow could be detected; 3 when very strong blood-flow signals were present.

All patients will undergo pre-operative MRI scan and PET/CT scan. Pelvic exenteration and laterally-extended pelvic resection will be performed with the aim to remove en bloc the recurrent or persistent disease with a free-of-tumor margin.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients with histologically-proven recurrent or persistent gynecological cancer who are planned to undergo pelvic exenteration or laterally extended pelvic resection, both with curative and with palliative intent.

* Anterior/total pelvic exenteration
* Laterally extended endopelvic resection (LEER)
* Laterally extended pelvic resection (LEPR) is defined as an en bloc lateral resection of a pelvic tumor involving sidewall muscle, and/or bone, and/or major nerve, and/or major vascular structure
* With or without stoma formation

Exclusion Criteria:

* Radical hysterectomy without lateral resection
* Rectal resection only (posterior exenteration)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing pelvic evisceration and lateral pelvic resection
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
pelvic exenteration resection. | 30 minutes
  The accuracy of US in the assessment of pelvic structures involvement in recurrent/persistent gynecologic tumors with disease limited to the pelvis.

SECONDARY OUTCOMES:
accuracy of US with the accuracy of MRI | 1 week
  To compare accuracy of US with the accuracy of MRI scan using histology as standard.

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIA CARLA TESTA, PROF, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT06278610/Prot_000.pdf